CLINICAL TRIAL: NCT02545309
Title: Secondary Sclerosing Cholangitis in Critically Ill Patients (SSC-CIP): A Pilot Study on the Possible Genetic Basis of the Disease
Brief Title: Secondary Sclerosing Cholangitis in Critically Ill Patients
Acronym: SSC-CIP
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 26-569 ex 13/14
Record Dates: First submitted 2015-07-29; First posted 2015-09-09 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Secondary Sclerosing Cholangitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum Stool Urine DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SSC-CIP: Patients with secondary sclerosing cholangitis in critically ill patients
- control: Patients with similar degree of critical illness who do not develop secondary sclerosing cholangitis in critically ill patients

SUMMARY:
SSC-CIP is increasing in patients after critical illness. Pathogenesis is still largely unclear. The investigators hypothesize that genetic variants of biliary transporter genes are frequent in patients with SSC-CIP. In approximately 140 patients and controls the rate of genetic variants in biliary transporter genes, gut permeability and gut microbiome as well as bone health will be studied.

DETAILED DESCRIPTION:
SSC is a process of fibroobliteration of intra- and extrahepatic bile ducts due to the fact that the bile ducts receive their blood supply exclusively through the hepatic artery and therefore are more prone to ischemia than other parts of the liver. Several factors, such as intraductal stone disease, surgical or blunt abdominal trauma, intra-arterial chemotherapy, and recurrent pancreatitis can lead to SSC. A relatively new entity is SSC occurring after critical illness (SSC-CIP). So far 97 cases have been reported in literature. All these patients recovered from critical illness, where they received ventilation with positive end-expiratory pressure and vasopressors. A rapid increase in cholestasis and irregular strictures of the intrahepatic bile ducts were observed within weeks after the onset of the critical illness. On endoscopic retrograde cholangiography typically biliary casts can be found. Patients with SSC-CIP furthermore have a distinct microbial profile in bile with frequent detection of difficult to treat organisms. To date, only liver transplantation (in selected patients) provides a curative treatment. Prognosis of SSC-CIP is poor with a mortality rate of 36% after 18 months and the need for liver transplantation in 23%.

To date not much is known about potential risk factors for the development of SSC-CIP. Since not all patients receiving high pressure ventilation and vasopressors develop SSC-CIP, it can be hypothesized that other, patient-specific, factors may play a role in the development of SSC-CIP. Since it is a disease of bile ducts, genetic variants in biliary transporters might play a role. Genetic variants of bile acid transporters, such as BSEP (Bile salt export pump) or MDR3 (multidrug resistance protein 3) have been described as inducers and modifiers of liver disease, such as intrahepatic cholestasis of pregnancy, drug induced cholestasis or treatment success of hepatitis C.

Another potentially important but underreported problem in SSC-CIP is impaired bone health. It is well known, that chronic liver disease, often results in metabolic bone disease: reduced bone mineral density is found in up to 60% and atraumatic fractures in 20% of patients. Specifically chronic cholestatic liver disease is associated with increased fracture risk. This can result in spontaneous or low-impact fractures in such patients, adversely affecting quality of life and survival.

However, no data on bone mineral density and bone mineral metabolism in SSC-CIP are available yet.

The investigators therefore aim to analyse a panel of potentially relevant genes in bile acid transport and bile composition in patients with SSC-CIP to identify potential genetic variants associated with the development of SSC-CIP. Serum markers of bone mineral metabolism and osteodensitometry data will be obtained too. Furthermore, since the microbial profile in bile of SSC-CIP patients shows a predominance of difficult to treat pathogens, changes in gut microbiome composition and/or gut permeability with consecutive translocation of bacterial products into the circulation might be of relevance. From a clinical point of view mortality in SSC-CIP is often related to multi-organ failure. Since infections play an important role in the development of multi-organ failure, the investigators also hypothesize, that SSC-CIP leads to an impairment of innate immune responses.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Age above 18 years
* secondary sclerosing cholangitis in critically ill patients

Exclusion Criteria:

* mechanical cholestasis
* primary sclerosing cholangitis
* primary biliary cirrhosis
* Immune globulin G4 associated cholangitis
* toxic cholestasis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with no liver disease in the past, who develop secondary sclerosing cholangitis during/after a critical illness
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2015-12-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
bile acid transporter genes | Day 1
  Rate of genetic variants in biliary transporter genes

SECONDARY OUTCOMES:
gut permeability | Day 1
  degree of increase in gut permeability
bile acids | Day 1
  changes in bile acid composition
bone health | Day 1
  Lumbar spine Z-Scores
upper gastrointestinal bleeding episodes | through study completion, an average of 3 years (from date of inclusion through end of observation/death)
  gastrointestinal bleeding on upper gastrointestinal endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria